CLINICAL TRIAL: NCT02264600
Title: Oxidative Stress and Apelin Level in Willis Ekbom Disease
Brief Title: Apelin in Willis Ekbom Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Selda Korkmaz, Principal Investigator, Acibadem University
Other Study IDs: AWED-31014
Record Dates: First submitted 2014-10-03; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome, Apelin, Oxidative Stress
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess apelin level in patients with Willis-Ekbom Disease (WED) as known Restless Legs Syndrome (RLS). Cardiovascular complications of WED have been reported in recent studies. Increased oxidative stress is thought to play an important role in cardiovascular complications of WED patients. Apelin is a novel described antioxidant bioactive peptide. The investigators hypothesize that patients with WED have lower plasma apelin level than healthy subjects based on presence of oxidative stress of WED.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as RLS/WED according to International Classification of Sleep Disorders (ICSD-3) criteria
* Patients with idiopathic RLS/WED
* Moderate and severe RLS/WED according to International Restless Legs Syndrome Rating Scale
* Periodic Leg Movements Index above 5 in polysomnography record
* BMI below 25

Exclusion Criteria:

* Disorders which cause symptomatic RLS(Iron deficiency anemia, kidney failure, diabetes mellitus, pregnancy, Parkinson's disease, multiple sclerosis, neuropathy)
* Systemic diseases which cause possible oxidative stress status (cardiovascular diseases, obesity, diabetes mellitus, use of any medical drugs especially ACE inhibitors e.g.)
* Another sleep disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who are administered to Kayseri Acibadem Hospital Sleep Medicine Unit, outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Serum apelin level in WED patients and healthy controls | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Murat Aksu, Prof. Dr., Study Director — Acibadem University Faculty of Medicine, School of Electroneurophysiology

REFERENCES:
- [Background] Cikrikcioglu MA, Hursitoglu M, Erkal H, Kinas BE, Sztajzel J, Cakirca M, Arslan AG, Erek A, Halac G, Tukek T. Oxidative stress and autonomic nervous system functions in restless legs syndrome. Eur J Clin Invest. 2011 Jul;41(7):734-42. doi: 10.1111/j.1365-2362.2010.02461.x. Epub 2011 Jan 20. PMID 21250984
- [Background] Baskol G, Korkmaz S, Erdem F, Caniklioglu A, Kocyigit M, Aksu M. Assessment of nitric oxide, advanced oxidation protein products, malondialdehyde, and thiol levels in patients with restless legs syndrome. Sleep Med. 2012 Apr;13(4):414-8. doi: 10.1016/j.sleep.2011.11.012. PMID 22469072
- [Background] Boucher J, Masri B, Daviaud D, Gesta S, Guigne C, Mazzucotelli A, Castan-Laurell I, Tack I, Knibiehler B, Carpene C, Audigier Y, Saulnier-Blache JS, Valet P. Apelin, a newly identified adipokine up-regulated by insulin and obesity. Endocrinology. 2005 Apr;146(4):1764-71. doi: 10.1210/en.2004-1427. Epub 2005 Jan 27. PMID 15677759
- [Background] Lv SY, Qin YJ, Wang HT, Xu N, Yang YJ, Chen Q. Centrally administered apelin-13 induces depression-like behavior in mice. Brain Res Bull. 2012 Sep 1;88(6):574-80. doi: 10.1016/j.brainresbull.2012.06.003. Epub 2012 Jun 21. PMID 22728209
- See also: Related Info — http://www.rls.org